CLINICAL TRIAL: NCT01596270
Title: A Phase 1 Dose-escalation Study of the Safety and Pharmacokinetics of a Tablet Formulation of SAR245409 Administered Daily to Patients With Solid Tumors or Lymphoma
Brief Title: A Study of the Safety and Pharmacokinetics of SAR245409 Tablets in Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TED12471; U1111-1123-1488 (Other: UTN)
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2014-10

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — XL765

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Once daily dosing (Experimental): escalating doses, once daily dosing every day, no eating for 2 hours prior and 1 hour after dose
  Interventions: Drug: SAR245409
- Twice daily dosing (Experimental): escalating doses, twice daily dosing every day, no eating for 2 hours prior and 1 hour after dose
  Interventions: Drug: SAR245409

INTERVENTIONS:
Drug: SAR245409 — Pharmaceutical form: tablet Route of administration: oral

SUMMARY:
Primary Objective:

- To evaluate the safety and tolerability of SAR245409 tablets administered once or twice a day in patients with solid tumors or lymphoma.

Secondary Objectives:

* To evaluate blood levels of SAR245409 after administration of SAR245409 tablets once or twice a day in patients with solid tumors or lymphoma.
* To evaluate the effect of food on blood levels of SAR245409 after administration of SAR245409 tablets in patients with solid tumors or lymphoma.
* To evaluate the effect of SAR245409 on the body after administration of SAR245409 tablets once or twice a day in patients with solid tumors or lymphoma.
* To obtain information on how SAR245409 administered once or twice a day to patients with solid tumors or lymphoma affect disease symptoms and study treatment side effects as reported by the patients on a questionnaire.
* To explore the antitumor activity of SAR245409 tablets administered once or twice a day to patients with solid tumors or lymphoma.

DETAILED DESCRIPTION:
The total study duration per patient will be 58 to 128 days and will include a screening period (1 to 28 days), a food interaction investigation period (when applicable; 4 to 11 days), two 28-day treatment cycles (56 days), an end-of-treatment visit (within 7 days after the last SAR245409 administration) and a follow-up visit (within 30 ± 3 days after the last SAR245409 administration).

ELIGIBILITY:
Inclusion criteria :

* Solid tumor that is metastatic or unresectable, or relapsed or refractory lymphoma (including chronic lymphocytic leukemia/small lymphocytic lymphoma), for which standard therapies are no longer effective or there are no therapies known to prolong survival.
* Male or female patient > or = 18 years old.
* Eastern Cooperative Oncology Group Performance Status < or = 1.
* Adequate white blood cells, platelets and haemoglobin.
* Adequate liver and kidney functions.
* Fasting plasma glucose < 160 mg/dL.
* No other malignancy.
* Women of childbearing potential using adequate contraception.

Exclusion criteria:

* History of partial or full gastrectomy.
* Lymphoma involving the gastrointestinal tract.
* Uncontrolled brain metastases or a primary brain tumor.
* Prior treatment with cytotoxic chemotherapy (including investigational agents) or biologic agents (antibodies, immune modulators, and cytokines) within 4 weeks, or nitrosoureas or mitomycin C within 6 weeks, before the first dose of study treatment.
* Prior treatment with a small-molecule kinase inhibitor (including investigational agents) within 2 weeks, or 5 half lives of the drug or active metabolites, whichever is longer, before the first dose of study treatment.
* Any other investigational therapy within 4 weeks before the first dose of study treatment.
* Prior anticancer hormonal therapy within 1 week before the first dose of study treatment.
* Prior radiation therapy within 2 weeks before the first dose of study treatment.
* Intolerance of prior treatment with a PI3K inhibitor.
* Hereditary or acquired immunodeficiency syndrome or HIV (human immunodeficiency virus) infection.
* Lymphoma patients with positive serologies for Hepatitis B surface antigen (HBsAg) or anti-Hepatitis C virus (anti-HCV) antibodies.
* Positive serologies for Hepatitis B surface antigen (HBsAg) or anti-Hepatitis C virus (anti-HCV) antibodies.
* Patient is pregnant or breastfeeding.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | Up to Day 28

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events | From first dose of SAR245409 until 30 days after the last dose
Maximum SAR245409 plasma concentration | Cycle 1 Days 1, 2, 8, 15, and 28, and Cycle 2 Day 1
Area under the SAR245409 plasma concentration versus time curve | Cycle 1 Days 1, 2, 8, 15, and 28, and Cycle 2 Day 1
Ratio of maximum SAR245409 plasma concentration between fed and fasted dosing | Days 1, 2, 3, and 4 of the food interaction period
Ratio of area under the SAR245409 plasma concentration versus time curve between fed and fasted dosing | Days 1, 2, 3, and 4 of the food interaction period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 840001, Detroit, Michigan
  - Investigational Site Number 840002, New Brunswick, New Jersey
  - Investigational Site Number 840003, Dallas, Texas